CLINICAL TRIAL: NCT03706391
Title: Study of ALS Reversals 4: LifeTime Exposures
Acronym: StARLiTE
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National ALS Registry (Unknown); Centers for Disease Control and Prevention (U.S. Federal Agency); Agency for Toxic Substances and Disease Registry (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00100219
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2020-07

CONDITIONS: Amyotrophic Lateral Sclerosis; Progressive Muscular Atrophy; Motor Neuron Disease
Keywords: amyotrophic lateral sclerosis; progressive muscular atrophy; motor neuron disease; ALS Reversal; PMA Reversal
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Muscular Atrophy, Spinal; Motor Neuron Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ALS and PMA Reversals

SUMMARY:
Hypothesis: There exists patients who have met ALS or PMA diagnostic criteria and subsequently experienced robust and sustained improvement, i.e. a "reversal." Thirty-eight of these patients were identified in the prior Duke University study, Documentation of Known ALS Reversals (St.A.R. Protocol 1, Duke IRB Pro00076395). The investigators hypothesize these patients have had different environmental exposures than patients with typically progressive ALS. Identification of specific environmental influences may point to exposures which are protective or exposure that lead to the development of a rare and novel reversible ALS-like disease.

Objective: This study seeks to identify environmental exposures associated with ALS reversals.

DETAILED DESCRIPTION:
Amyotrophic Lateral Sclerosis (ALS) is a devastating motor neuron disease that typically causes rapidly progressive muscle weakness, disability and premature death. In spite of a large number of attempted ALS trials, there are no significant disease-modifying therapies for this condition to-date.

There exists a small group of patients who meet diagnostic criteria for ALS or progressive muscular atrophy (PMA), progress for a period of time, and then significantly improve. Some of these "ALS reversals" even make a complete recovery back to normal neurological function. The investigators have independently verified 38 of these cases so far through review of medical records and peer-reviewed literature. These patients are different in their demographics and disease characteristics as compared to patients with more typically progressive ALS.

One possible explanation for these cases is that these patients have had protective environmental exposures. Another possible explanation is that these patients have had unique environmental exposures that led to a reversible form of ALS. Study of these selected reversal patients may yield valuable clues to environmental mechanisms of ALS resistance.

This is a pilot case-control study attempting to discover environmental exposure correlates to ALS reversals. The investigators will recruit and enroll ALS reversal "cases" to fill out an online survey form about their life. Topics include demographics, employment history, military service, substance use, physical activity, family medical history, disease progression, residential history, occupational exposures, home exposures, hobby exposures, hormonal and reproductive history (female identifying subjects only), caffeine, head and neck injuries, electrical shocks, health insurance, subjective perception of the etiology of ALS, and clinical features of disease. "Control" participant data will come from a pre-existing database.

ELIGIBILITY:
Inclusion Criteria:

* Prior participation in Documentation of Known ALS Reversals (Duke IRB Pro00076395)
* Confirmation of ALS or PMA (primary muscular atrophy) diagnosis through medical record review (previously documented in Documentation of Known ALS Reversals protocol)
* Sustained, robust improvement on at least one objective ALS outcomes measure (ex. ALSFRS-R, FVC, strength testing, EMG) (previously documented in Documentation of Known ALS Reversals protocol)
* Able to understand English

Exclusion Criteria:

* History of cognitive impairment severe enough to preclude informed consent, reported by patient on direct questioning or as suspected by research personnel from Documentation of Known ALS Reversals (Duke IRB Pro00076395) study data

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from the cohort of subjects (38 to-date) who participated in the Documentation of Known ALS Reversals (Duke IRB Pro00076395) protocol and were subsequently thought to have an ALS Reversal.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Life Time Environmental Exposures | 2 hours to fill out survey
  Case-control analysis of differences in environmental exposures over life time of subject. Environmental exposures will be measured with the National ALS Registry survey. Cases are "ALS Reversals." Controls are typically progressive patients with ALS.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke ALS Clinic / DUSOM Dept of Neurology / DUHS, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ALSUntangled Group. ALSUntangled No. 12: Dean Kraft, Energy Healer. Amyotroph Lateral Scler. 2011 Sep;12(5):389-91. doi: 10.3109/17482968.2011.609309. No abstract available. PMID 21981685
- [Background] Bedlack RS, Vaughan T, Wicks P, Heywood J, Sinani E, Selsov R, Macklin EA, Schoenfeld D, Cudkowicz M, Sherman A. How common are ALS plateaus and reversals? Neurology. 2016 Mar 1;86(9):808-12. doi: 10.1212/WNL.0000000000002251. Epub 2015 Dec 9. PMID 26658909
- [Background] http://www.wsj.com/articles/the-mystery-of-als-patients-who-see-improvement-1465845332
- [Background] Harrison D, Mehta P, van Es MA, Stommel E, Drory VE, Nefussy B, van den Berg LH, Crayle J, Bedlack R; Pooled Resource Open-Access ALS Clinical Trials Consortium. "ALS reversals": demographics, disease characteristics, treatments, and co-morbidities. Amyotroph Lateral Scler Frontotemporal Degener. 2018 Nov;19(7-8):495-499. doi: 10.1080/21678421.2018.1457059. Epub 2018 Apr 2. PMID 29607695
- [Background] Crayle J and Bedlack R. Unpublished data. 2018.